CLINICAL TRIAL: NCT02438085
Title: Acute coRonary sYndrOmes proSpective regisTry Of Ferrara
Brief Title: Prospective Registry of Acute Coronary Syndromes in Ferrara
Acronym: ARYOSTO
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Assistant Professor and Interventional Cardiologist, University Hospital of Ferrara
Other Study IDs: 073132
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Acute Coronary Syndromes
Keywords: acute coronary syndromes; outcome; medical management; comorbidities; registry
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — whole blood, plasma, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ACS patients: prospective collection of data and follow-up
  Interventions: Other: prospective collection of data and follow-up

INTERVENTIONS:
Other: prospective collection of data and follow-up — prospective collection of data and follow-up of all patients admitted to hospital for ACS

SUMMARY:
The ARYOSTO has been designed to describe the clinical epidemiology and the current management of acute coronary syndromes (ACS) in the area of Ferrara. Especially, the Authors will evaluate the medical and interventional management of ACS patients admitted to hospitals in the area of Ferrara and receiving coronary artery angiography and percutaneous coronary intervention (PCI) in the hub center of Ferrara (Azienda Ospedaliera Universitaria di Ferrara, Cona (FE), Italy)

DETAILED DESCRIPTION:
The Cardiovascular Institute of the University Hospital of Ferrara is the hub center of the area of Ferrara (400.000 residents). The cath-lab of the University Hospital of Ferrara is the hub center of the network for the management of patients with ACS. This finding guarantees a very high number of patients with ACS admitted to University Hospital of Ferrara (more than 1500 by year). In the cath-lab are performed more than 2000 coronary artery angiography by year and more than 1100 PCI by year. The staff of the cardiology unit has a great experience in the management of studies (investigator-driven, randomized controlled trials, with or without sponsor) enrolling patients with ACS and treated with PCI. All consecutive patients with ACS admitted to hospitals of the Ferrara area will be included in the registry. All data will be related to long-term clinical outcome.

METHODS:

Prospective collection of following data:

* baseline characteristics including cardiovascular (CV) risk factors, CV history and comorbidities (see below)
* clinical management (CV drugs, imaging exams, diagnostic exams, time to cath-lab access)
* biomarkers evaluating inflammation, endothelial, platelet, thrombotic function and activation
* procedural details including coronary disease description, intervention modality, stent, coronary imaging, CV drugs during intervention, procedural complications and management, access site
* in-hospital adverse events
* medical treatment at discharge and during the follow-up
* clinical follow-up (1, 2, 3, 4 5 years)

PRE-SPECIFIED SUBSTUDY

The Authors will focus the attention in specific subset of patients:

* patients with diabetes
* patients with chronic obstructive pulmonary disease
* patients with chronic kidney disease
* patients with rheumatologic disordes
* patients with malignancy In these subsets of patients the Authors will collect a more detailed description of symptoms, clinical presentation, disease management and relationship between comorbidity and ACS.

Similarly, a specifc substudy of the registry will be focused on the characterization of coronary artery disease and of atherosclerotic plaque morphology in patients with comorbidities (diabetes, COPD, CKD, malignancy) as compared to patients without comorbidities.

Finally, the Authors will evaluate the quality of life of ACS patients in the area of Ferrara applying at 1, 2, 3, 4 and 5 years the following questionnaires: EQ-5D and SF-12 v2

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* hospital admission for acute coronary syndromes
* resident in the Ferrara area

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to hospital with diagnosis of acute coronary syndromes according current European guidelines
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
1-year combined primary endpoint | 1 year
  1-year occurence of cardiac death, myocardial infarction, cerebrovascular accident

SECONDARY OUTCOMES:
2-year combined endpoint | 2 years
  2-year occurence of cardiac death, myocardial infarction, cerebrovascular accident
3-year combined endpoint | 3 years
  3-year occurence of cardiac death, myocardial infarction, cerebrovascular accident
5-year combined endpoint | 5 years
  5-year occurence of cardiac death, myocardial infarction, cerebrovascular accident
annual occurrence of single components of primary endpoint | 1, 2, 3, 4, 5 years
  occurrence of each component of the primary endpoint
primary safety outcome | 1 year
  1 year occurrence of BARC 2-3 bleedings
cardiac adverse events | 1, 2, 3, 4, 5 years
  hospital admission heart failure, arrhytmias, acute coronary syndromes, admission to emergency room for chest pain
respiratory adverse events | 1, 2, 3, 4, 5 years
  hospital admission for respiratory cause

OTHER OUTCOMES:
emergency room admittance | 1, 2, 3, 4, 5 years
  assessment of number of admission to emergency room for any causes

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

REFERENCES:
- [Derived] Cimaglia P, Fortini F, Vieceli Dalla Sega F, Cardelli LS, Massafra RF, Morelli C, Trichilo M, Ferrari R, Rizzo P, Campo G. Relationship between PCSK9 and endothelial function in patients with acute myocardial infarction. Nutr Metab Cardiovasc Dis. 2022 Sep;32(9):2105-2111. doi: 10.1016/j.numecd.2022.06.020. Epub 2022 Jul 2. PMID 35915019
- [Derived] Pavasini R, Fabbri G, Marchini F, Bianchi N, Deserio MA, Sanguettoli F, Verardi FM, Segala D, Pompei G, Tonet E, Serenelli M, Caglioni S, Guardigli G, Campo G, Cultrera R. Procalcitonin Predicts Bacterial Infection, but Not Long-Term Occurrence of Adverse Events in Patients with Acute Coronary Syndrome. J Clin Med. 2022 Jan 22;11(3):554. doi: 10.3390/jcm11030554. PMID 35160005